CLINICAL TRIAL: NCT06645444
Title: Immediate Implant Placement With Different Materials of Customized Healing Abutment for Guiding Peri-implant Soft Tissue Healing in Posterior Teeth: A Randomized Controlled Clinical Trial
Brief Title: Immediate Implant Placement With Different Materials of Customized Healing Abutment for Guiding Peri-implant Soft Tissue Healing in Posterior Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Helal, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 591024
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant placement with customized composite healing abutment (Active Comparator): * extraction of the Posterior teeth will be done with minimally invasive technique using periotome.
  * Then, the digital surgical guide will be placed, and will be checked the affinity of the reference window with other teeth accurately in the optimal position. The osteotomies will be prepared with a surgical-guided surgery kit through a digital surgical guide and drill direction will be ensured by radiographic taking. Implant fixture insertion will be performed through this digital surgical guide.
  * All patients will receive a bone-level implant with varying diameter and length in each case. After implant placement, the operator will scan the surrounding gingiva with a scan body immediately for a post-extraction digital model.
  * Then the spaces between the implant fixture and alveolar bone wall will be filled with locally harvested autogenous bone and xenograft grafting material (OsteoBiol Gen-Os, Sweden).
  Interventions: Other: immediate implant placement with customized PEEK healing abutment
- immediate implant placement with customized PEEK healing abutment (Experimental): * an intraoral examination will be done and a digital impression will be taken by the intraoral scanner (MEDIT i500) for a pre-extraction digital model, and CBCT will be taken for prosthetic-driven planning.
  * Once the treatment plan formulated, both STL (Standard Triangle Language) and DICOM (CBCT raw data) files format will be sent to produce the digital surgical guide with metal sleeve.
  * Then, a customized PEEK healing abutment will be made mimicking the anatomical cervical contour and pseudo-CEJ will be made by merging the STL and DICOM digitally and the exterior surface of the healing abutment will be designed to resemble a tooth.
  * Then, the technicians will mill the customized healing abutment digital design from a pre-milled 14 × 14 mm PEEK block (BioHPP, Bredent®, Bolzano, Italy) with a non-hex connection type, polished it, and sterilized it.
  * The digital surgical guide with a metal sleeve will be back for scheduled patient implant surgery.
  Interventions: Other: immediate implant placement with customized PEEK healing abutment

INTERVENTIONS:
Other: immediate implant placement with customized PEEK healing abutment — * an intraoral examination will be done and a digital impression will be taken by the intraoral scanner (MEDIT i500) for a pre-extraction digital model, and CBCT will be taken for prosthetic-driven planning.
  * Once the treatment plan formulated, both STL (Standard Triangle Language) and DICOM (CBCT raw data) files format will be sent to produce the digital surgical guide with metal sleeve.
  * Then, a customized PEEK healing abutment will be made mimicking the anatomical cervical contour and pseudo-CEJ will be made by merging the STL and DICOM digitally and the exterior surface of the healing abutment will be designed to resemble a tooth.
  * Then, the technicians will mill the customized healing abutment digital design from a pre-milled 14 × 14 mm PEEK block (BioHPP, Bredent®, Bolzano, Italy) with a non-hex connection type, polished it, and sterilized it.
  * The digital surgical guide with a metal sleeve will be back for scheduled patient implant surgery.

SUMMARY:
: Immediate Implant Placement with different materials of customized healing abutment for guiding Peri-implant Soft Tissue Healing in Posterior Teeth: A Randomized controlled clinical trial.

DETAILED DESCRIPTION:
This randomized clinical trial evaluates the effect of customized PEEK healing abutment versus composite healing abutment regarding Clinical evaluation

1. Gingival margin distance
2. Gingival margin height
3. Gingival contour width
4. Gingival volume in BL & MD aspects on guiding the peri- implant soft tissue emergency profile in posterior teeth after immediate implant placement

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria of participants:

  * Periodontally and systemic healthy patients
  * Patients aged > 18 years
  * Non- restored teeth for many reasons (i.e. endodontic failure, unworthy for treatment in deep caries/non-caries lesion and root fracture), locate in the posterior area in the maxillary or mandibular arch indicate for customized implant with no need for additional bone and soft tissue augmentation procedures.
  * An adequate vertical bone for immediate implant placement.
  * Implants will be positioned with adequate primary stability so that transmucosal healing can be accomplished.
  * No taken medications known to interfere healing or periodontal tissue health or bone metabolism.
  * No previous periodontal surgery at involved sites.
  * Good oral hygiene and good compliance with the plaque control instructions following initial therapy.

Exclusion criteria:

* Patients with active periodontal diseases (bleeding on probing- probing depth > 4 mm) or those under orthodontic treatment.
* Poor oral hygiene (full mouth plaque score > 25% and full mouth bleeding score > 25%)
* Smoking habits (> 10 cigarettes/day)
* Severe acute or chronic periodontitis
* Severe bruxism habits
* History of oral/IV bisphosphonates taking
* Remote or recent radiation therapy in the oro-maxillo-facial area or recent chemotherapy.
* Xerostomia
* Pregnant and lactating mothers
* Patients who have been received periodontal surgery in the study area during the last year.
* Clinical or radiographic signs of periapical pathology contraindicating immediate implant placement.
* Implants showing signs of peri-implant mucositis and peri-implantitis during the study period will be excluded from the following analyses.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Gingival margin distance | Day 0 - month 3
  The gingival margin distance will be measured from the highest gingival margin point in the buccal, palatal/lingual, mesial, and distal sides to the longitudinal implant line parallelly with the platform plane (buccal margin distance; BD, palatal/lingual margin distance; LD, mesial margin distance; MD and distal margin distance; DD).
Gingival margin height | Day 0 - month 3
  Gingival margin height will be measured from the highest gingival margin point in the buccal, lingual, mesial, and distal sides perpendicular to the platform plane (buccal height; BH, palatal/lingual height; LH, mesial height; MH and distal height; DH).
Gingival contour width | Day 0 - month 3
  The contour width will be measured from the outer sur face on the buccal and lingual sides to the implant center on the platform plane (buccal width; BW and palatal/lingual width; LW).
Gingival volume in BL & MD aspects | Day 0 - month 3
  Gingival volume will be measured on the gingiva above the platform plane for total gingival volume and separated with a mid-mesiodistal plane through the implant center for buccal and lingual gingival volume (total buccolingual volume; BLV, buccal volume; BV and lingual volume; LV).

SECONDARY OUTCOMES:
The Functional Implant Prosthodontics Score | Day 0 - month 3
  The Functional Implant Prosthodontics Score will be measured through five variables in order to limit bias: (1) interproximal contact and papillae, (2) occlusion static and dynamic, (3) design color and contour, (4) mucosa quality and quantity, and (5) bone x-ray. A scoring scheme of 0-1-2 resulting in a maximum score of ten (5X2) per implant reconstruction.

OTHER OUTCOMES:
Numerical rating scale | Day 0 - 2 hours- 24 hours
  is a psychometric response to pain scale which will be used in questionnaires through asking the patients about the occurrence of discomfort and postoperative pain Will be evaluated by questionnaire to assess perceived pain following crown insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Helal, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3- months